CLINICAL TRIAL: NCT00292435
Title: A 12-week, Double-blind, Randomised, Placebo-controlled, Multicentre Trial to Evaluate Efficacy and Tolerability of Antistax Film-coated Tablets, 360 mg/Day Orally, in Male and Female Patients Suffering From Chronic Venous Insufficiency.
Brief Title: Efficacy and Tolerability CVI (A 12-week, Double-blind, Randomised, Placebo-controlled, Multicentre Trial (CVI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1138.10
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — AS 195

INTERVENTIONS:
Drug: Read vine leaf extract (AS 195)

SUMMARY:
To determine efficacy and tolerability of Antistax 360 mg tablets in chronic venous insufficiency linked to edema (swelling) and subjective symptoms

Age Groups: Child, Adult, Older Adult
Enrollment: 202
Dates: Start 2006-03; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in limb volume of the more affected leg on day 84 , determined by water displacement. | 84 days

SECONDARY OUTCOMES:
Change from baseline in limb volume on days 21 and 42 determined by water displacement. | 21 and 42 days
Change from baseline in calf circumference on days 21, 42, and 84 | 21, 42 and 84 days
Change from baseline in the subjective symptoms of CVI (tired heavy legs, sensation of tension in the legs, tingling sensations in the legs, pain in the legs) measured by visual analogue scales (VAS) on days 21, 42, and 84 | 21, 42 and 84 days
Global assessment of efficacy by the patient on day 84 | 84 days
Global assessment of efficacy by the investigator on day 84 | 84 days
Change from baseline in quality of life as determined by the Tuebingen QoL Questionnaire on day 84 | 84 days
Incidence of adverse events | 84 days
Measurement of vital signs (pulse rate, blood pressure) | 84 days
Global assessment of tolerability by the patient and by the investigator on day 84. | day 84

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (16):
- Austria (3):
  - LKH Graz, Graz
  - AKH Wien, Vienna
  - VENEX Venenexperten, Vienna
- Czechia (2):
  - Boehringer Ingelheim Investigational Site, Brno
  - Neurology-geriatric Institute, Moravský Beroun
- Germany (11):
  - Boehringer Ingelheim Investigational Site, Berlin
  - Klinik und Poliklinik der Universitat Bonn, Bonn
  - Boehringer Ingelheim Investigational Site, Cologne
  - Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - Klinik und Poliklinik fur Hautkrankheiten, Greifswald
  - Klinikum der Johannes Gutenberg-Universitat, Mainz
  - Gesundheitszentrum Minden, Minden
  - Boehringer Ingelheim Investigational Site, München
  - Boehringer Ingelheim Investigational Site, Oberkirch
  - Boehringer Ingelheim Investigational Site, Rottweil
  - Universitats-Hautklinik, Tübingen